CLINICAL TRIAL: NCT01269892
Title: Study of Nutritional Regime for Acute Diarrhea
Brief Title: Early Administration of Lactose-free Milk in Children Presenting With Acute Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy, Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ASD-1213-9
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2009-01

CONDITIONS: Acute Diarrhea
Keywords: diarrhea, lactose, milk, weight, acute.
MeSH Terms: conditions — Diarrhea; Body Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lactose-free milk (Other): it is kind of nutritional regime
  Interventions: Dietary Supplement: lactose-free milk
- conventional milk (Other): it is kind of nutritional regime
  Interventions: Dietary Supplement: conventional milk

INTERVENTIONS:
Dietary Supplement: lactose-free milk — a milk without lactose
  Other Names: nothing
  Arms: lactose-free milk
Dietary Supplement: conventional milk — a milk with lactose
  Other Names: nothing
  Arms: conventional milk

SUMMARY:
The purpose of this study is to determine which nutritional regime is better for acute diarrhea in outcomes.

DETAILED DESCRIPTION:
Diarrhea is still the most important cause of mortality and morbidity in children of the developing countries. We evaluated the effectiveness of early administration of lactose free milk in the management of acute diarrhea in children below two years old.

ELIGIBILITY:
Inclusion Criteria:

1. children with acute non-bloody diarrhea (≤ 2 weeks)
2. mild to moderate dehydration

Exclusion Criteria:

1. mucous bloody stools
2. major systemic illness
3. severe malnutrition (Weight for age <60% and Weight for height <70 %)
4. history of antibiotics receiving

Ages: 3 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
duration of diarrhea | at seven days after admission
  Duration of diarrhea corresponded to the time from enrollment to the cessation of diarrhea, which was defined as the passage of the last watery or loose stool before passage of two consecutive formed stools or no stool in a 24-hour period.

SECONDARY OUTCOMES:
changes in weight gaining | at seven days after admission
  nude weight was measured with scale with an accuracy of 10 g at admission time and seven days after admission

CONTACTS AND LOCATIONS:
Overall Officials: Ali Gholamrezaei, MD, Study Chair — MD,research comittee
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran